CLINICAL TRIAL: NCT02781493
Title: Efficacy of Prucalopride Plus Polyethylene Glycol in Bowel Preparation for Colonoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Binzhou People's Hospital (Other); Tai'an People's Hospital (Unknown); Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016SDU-QILU-06
Record Dates: First submitted 2016-05-21; First posted 2016-05-24 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Prucalopride Plus Polyethylene Glycol in Bowel Preparation for Colonoscopyp
Keywords: Prucalopride; Polyethylene Glycol; bowel preparation
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prucalopride group (Experimental): 2 mg Prucalopride plus 2 L Polyethylene Glycol regimen
  Interventions: Drug: 2 mg Prucalopride plus 2 L Polyethylene Glycol regimen
- Placebo group (Placebo Comparator): 2 mg Placebo plus 2 L Polyethylene Glycol regimen
  Interventions: Drug: 2 mg Placebo plus 2 L Polyethylene Glycol regimen

INTERVENTIONS:
Drug: 2 mg Prucalopride plus 2 L Polyethylene Glycol regimen — Patients enrolled in the Prucalopride group will recieve 2 mg Linaclotide plus 2 L Polyethylene Glycol regimen before colonoscopy.
  Arms: Prucalopride group
Drug: 2 mg Placebo plus 2 L Polyethylene Glycol regimen — Patients enrolled in the Placebo group will recieve 2 mg Placebo plus 2 L Polyethylene Glycol regimen before colonoscopy.
  Arms: Placebo group

SUMMARY:
Prucalopride based bowel cleansing regimen might be helpful to improve bowel cleansing quality before colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is the standard approach for evaluating the colon currently. Thorough bowel cleansing is critical for adequate visualization of colonic mucosa during colonoscopy. Inadequate bowel cleansing results in adverse consequences for the examination, including lower adenoma detection rates, longer procedural time, lower cecal intubation rates, shorter intervals between examinations and an estimated 12-22% increase in overall colonoscopy cost.Unfortunately, despite advances in bowel preparation methods, up to one-third of all colonoscopies are reported to have an inadequate bowel preparation.

Prucalopride can accelerate colonic transit and has been demonstrated to be efficient in constipation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older,
* scheduled to undergo elective outpatient colonoscopy,
* and were able to provide informed consent.

Exclusion Criteria:

* history of colorectal surgery
* severe colonic stricture or obstructing tumour
* dysphagia
* compromised swallowing reflex or mental status
* significant gastroparesis or gastric outlet obstruction
* known or suspected bowel obstruction or perforation
* severe chronic renal failure (creatinine clearance<30 ml/min
* severe congestive heart failure (New York Heart Association class III or IV)
* uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* dehydration
* disturbance of electrolytes
* pregnancy or lactation
* haemodynamically unstable
* unable to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Difference of scores rating by Boston Bowel Preparation Scale between 2 groups. | 9 months
  This is an established rating scale to evaluate the quality of bowel prep. The ratings will be compared between 2 groups.

SECONDARY OUTCOMES:
Polyp detection rate between 2 groups. | 9 months
rate of adverse events between 2 groups. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China